CLINICAL TRIAL: NCT07088627
Title: Performance and Hormonal Responses to Different Training Modalities in Young Weightlifters: A Randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Bekir Tokay, Lecturer, PhD, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 07
Record Dates: First submitted 2025-07-18; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Weightlifting; Hormone; Young; Performance; Anaerobic Power; Strength Training Effects
Keywords: hormone levels; strength training methods; performance; weightlifting

STUDY DESIGN:
Intervention Model Description: This study uses a randomized parallel group design where participants are assigned to one of four groups: UG, SG, MG, or CG. Each group undergoes a distinct training intervention over eight weeks. The groups are assessed pre- and post-intervention to evaluate differences in weightlifting performance, anaerobic power, and hormonal responses. The study aims to compare the effects of different strength training protocols on young male weightlifters while maintaining group homogeneity through stratified randomization and blinding of performance testers.
Who Masked: Outcomes Assessor
Masking Description: Only the individuals conducting performance assessments and hormone analyses were blinded to group assignments to minimize bias. No other parties were masked in this trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1: Undulating Strength Training Group (UG) (Experimental): Participants in this group follow an undulating periodization strength training protocol focused on the SN and C&J exercises. Training variables such as intensity (approximately 80% of 1RM) and volume (5 sets with descending repetitions: 5, 4, 3, 2, 1) vary weekly to stimulate neuromuscular adaptations. Rest intervals between sets are standardized at 90 seconds to optimize recovery and training quality.
  Interventions: Procedure: Intervention 1: UG
- Arm 2: Serial Strength Training Group (SG) (Experimental): Participants perform a serial strength training program emphasizing the SN and C&J exercises, with consistent load progression at approximately 80% of 1RM and a fixed volume of 5 sets of 5 repetitions per session. Rest periods between sets are set at 90 seconds to maintain training intensity and facilitate strength gains.
  Interventions: Procedure: Intervention 2: SG
- Arm 3: Maximal Strength Training Group (MG) (Experimental): This group engages in maximal strength training focused on high-intensity loads (around 100% of 1RM) with low volume (5 sets of 1 repetition) for SN and C&J exercises. Longer rest intervals of 180 seconds between sets are implemented to ensure adequate recovery for maximal effort lifts and to optimize peak strength development.
  Interventions: Procedure: Intervention 3: MG
- Arm 4: Control Group (CG) (No Intervention): Participants maintained their regular weightlifting routines, including the SN and C&J, without any additional intervention. Typical training loads range between 80-100% 1RM, with volume between 1 to 5 sets of 1 to 3 repetitions, without progressive overload or structured periodization. Rest intervals average 120 seconds between sets.

INTERVENTIONS:
Procedure: Intervention 1: UG — Participants perform UG targeting SN and C&J exercises, varying intensity at 80% of 1RM and volume (5 sets of 5, 4, 3, 2, 1 repetitions) over weeks. Rest between sets: 90 seconds.
  Arms: Arm 1: Undulating Strength Training Group (UG)
Procedure: Intervention 2: SG — Participants perform SG with SN and C&J at consistent 80% 1RM intensity, 5 sets of 5 repetitions each session. Rest between sets: 90 seconds.
  Arms: Arm 2: Serial Strength Training Group (SG)
Procedure: Intervention 3: MG — Participants engage in MG training focusing on SN and C&J at 100% 1RM, 5 sets of 1 repetition, with 180 seconds rest between sets.
  Arms: Arm 3: Maximal Strength Training Group (MG)

SUMMARY:
Olympic weightlifting is a sport that requires high levels of force production, technical skill, and intermuscular coordination. The effects of strength training during adolescence on performance, anaerobic power, and hormonal responses are critically important for athlete health and development.

This study investigated the effects of different strength training methods on snatch (SN) and clean & jerk (C&J) performance, anaerobic power levels, and selected hormonal parameters (growth hormone (GH), insulin-like growth factor 1 [IGF-1], total testosterone (TT), insulin (INS), thyroid-stimulating hormone (TSH)) in young male weightlifters. A total of 32 male weightlifters participated in the study. The participants were randomly assigned to one of four groups: undulating strength training (UG) (age: 17.6 ± 1.6 years), serial strength training (SG) (age: 16.9 ± 1.3 years), maximal strength training (MG) (age: 17.3 ± 1.4 years), and a control group (CG) (age: 17.1 ± 1.2 years). The experimental groups underwent sport-specific strength training five days per week for eight weeks. The performance assessments included one-repetition maximum (1RM) tests for the SN and C&J lifts, whereas the anaerobic power was measured via the vertical jump test. Hormonal parameters were analyzed via a chemiluminescent autoanalyzer. Paired samples t tests were used for within-group comparisons, and one-way analysis of variance (ANOVA) was employed for between-group comparisons.

The findings revealed significant improvements in SN, C&J, and anaerobic power performance in the groups subjected to UG, SG, and MG strength training. However, no significant differences were observed between the training groups in terms of performance or hormonal response. While some hormonal parameters increased, others did not significantly change.

Various strength training approaches contribute to improvements in the technical performance and anaerobic power of young weightlifters; however, their effects on hormonal responses appear to be limited. Planning training programs according to individual needs and developmental stages is essential for safeguarding athlete health and supporting long-term performance development.

DETAILED DESCRIPTION:
This experimental study examined the effects of three different strength training methods-undulating, serial, and maximal-on Olympic weightlifting performance, anaerobic power, and hormonal responses in adolescent male athletes. A total of 32 licensed male weightlifters with similar training backgrounds and weight categories were randomly assigned to four groups using stratified randomization. To maintain internal validity, group allocation was based on baseline metrics including age, training history, body weight, and performance measures.

The 8-week training intervention was delivered five days per week, with standardized session structures and rest intervals tailored to each protocol's physiological goals. Training programs targeted the SN and C&J exercises and were adjusted weekly based on reassessed one-repetition maximum (1RM) values. All sessions were conducted under the supervision of certified coaches to ensure technical consistency.

Anaerobic power was assessed using vertical jump tests, and hormonal measurements (GH, IGF-1, TT, INS and TSH) were obtained through venous blood samples analyzed via chemiluminescence autoanalyzers. To reduce variability, all blood samples were collected in a fasted state at the same time of day before and after the training period.

Blinded testers conducted all performance assessments, and standard operating procedures were applied to enhance reliability. Data were analyzed using parametric statistical tests (paired t-tests, ANOVA with Tukey post hoc analysis) to evaluate within- and between-group differences.

The study received ethical approval from the Non-Interventional Clinical Research Ethics Committee of the Faculty of Sport Sciences at Selçuk University (Decision No: 07, Date: 28.01.2021). Written informed consent was obtained from all participants, and confidentiality was strictly maintained throughout the research process.

ELIGIBILITY:
Inclusion Criteria:

* Male sex
* At least three years of licensed weightlifting experience
* No serious musculoskeletal injuries in the past year
* No use of medications, hormones, or supplements during the study
* Voluntary participation with signed informed consent

Exclusion Criteria:

* Participants outside the specified age range or with noncompliance to inclusion criteria

Ages: 15 Years to 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — This study is intended exclusively for male participants. Only biologically male individuals are eligible for participation.
Enrollment: 32 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2022-08-03 (Actual)

PRIMARY OUTCOMES:
1. SN Performance | Baseline (Week 0) and Post-Intervention (Week 8)
  SN performance is assessed by the maximum weight (in kilograms) successfully lifted in a 1RM test, recorded according to official International Weightlifting Federation (IWF) standards. The direction of improvement is indicated by an increase in lifted weight (kg).
2. C&J Performance | Baseline (Week 0) and Post-Intervention (Week 8)
  C&J performance is assessed by the maximum weight (in kilograms) successfully lifted in a 1RM test according to IWF standards. The direction of improvement is indicated by an increase in lifted weight (kg).
3. Anaerobic Power Performance | Baseline (Week 0) and Post-Intervention (Week 8)
  Anaerobic power is estimated using the Sayers equation, calculated from vertical jump height and body weight:
  Anaerobic Power (Watts) = (60.7 × jump height [cm]) + (45.3 × body weight [kg]) - 2055 Higher watt values indicate greater anaerobic power output.

SECONDARY OUTCOMES:
1. Serum GH Level | Baseline and 24 hours post-final training session
  Venous blood samples were collected between 08:00-09:00 following an overnight fast, both prior to the first training session and 24 hours after the final session. Serum GH levels (ng/mL) were analyzed using chemiluminescence-based autoanalyzers (Roche Elecsys 2010) in a certified laboratory, known for their high sensitivity and specificity. Each sample was measured twice, and the highest value was recorded. An increase or modulation in GH levels was considered indicative of endocrine adaptation.
2. Serum IGF-1 Level | Baseline and 24 hours post-final training session
  Venous blood samples were collected and processed in the same manner as for GH-between 08:00-09:00 following an overnight fast, prior to the first and 24 hours after the final training session. Serum IGF-1 levels (ng/mL) were measured using chemiluminescence-based autoanalyzers (Roche Elecsys 2010) in a certified laboratory. Each sample was analyzed twice, and the highest value was recorded. An increase in IGF-1 level was interpreted as an indication of anabolic response.
3. Serum TT Level | Baseline and 24 hours post-final training session
  TT levels were measured from venous serum samples collected under the same standardized conditions-between 08:00-09:00 following an overnight fast, prior to the first and 24 hours after the final training session. Measurements were performed using high-sensitivity chemiluminescence-based autoanalyzers (Roche Elecsys 2010) in a certified laboratory. Each sample was analyzed twice, and the highest value was recorded. An increase in testosterone levels was considered indicative of anabolic adaptation.
4. Serum INS Level | Baseline and 24 hours post-final training session
  INS concentration in serum was measured using the Roche Elecsys 2010 autoanalyzer following the same protocol-venous blood samples collected between 08:00-09:00 after an overnight fast, before the first and 24 hours after the final training session. Each sample was analyzed twice, and the highest value was used. Changes in insulin levels were interpreted as reflecting metabolic adjustment.
5. Serum TSH Level | Baseline and 24 hours post-final training session
  TSH levels were determined using certified chemiluminescence-based analysis. Venous blood samples were collected between 08:00-09:00 following an overnight fast, both before the first and 24 hours after the final training session. Each sample was measured twice, with the highest value recorded. Changes in TSH levels were interpreted as the thyroid regulatory hormone response to training stress.

CONTACTS AND LOCATIONS:
Overall Officials: Alpaslan Görücü, Professor Doctor, Study Director — Selçuk University, Faculty of Sport Sciences
Locations (1):
- Selçuk University, Faculty of Sport Sciences, Konya, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to ethical considerations and participant confidentiality constraints.